CLINICAL TRIAL: NCT02938949
Title: Alirocumab in Patients With Acute Myocardial Infarction: A Randomized Controlled Double-Blinded Study
Brief Title: Alirocumab in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20008008
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction; Hypercholesterolemia
Keywords: Myocardial Infarction; Low Density Lipoprotein Cholesterol; proprotein convertase subtilisin kexin 9, human; alirocumab
MeSH Terms: conditions — Myocardial Infarction; Hypercholesterolemia; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alirocumab (Active Comparator): Alirocumab (150 mg) will be administered by subcutaneous injection once, within the first day of the patient's diagnosis of NSTEMI. Patients will also receive an 80 mg dose of atorvastatin.
  Interventions: Drug: alirocumab
- placebo (Placebo Comparator): Placebo (sterile saline) will be administered by subcutaneous injection once, within the first day of the patient's diagnosis of NSTEMI. Patients will also receive an 80 mg dose of atorvastatin.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: alirocumab
  Other Names: Praluent
  Arms: Alirocumab
Drug: placebo
  Arms: placebo

SUMMARY:
Phase IV investigator initiated clinical trial to study the effectiveness of alirocumab, an inhibitor of proprotein convertase subtilisin/kexin (PCSK9), versus placebo added to high-intensity statin (atorvastatin 80 mg) in lowering low density lipoprotein (LDL) cholesterol during non-ST segment elevation myocardial infarction (NSTEMI).

DETAILED DESCRIPTION:
This research will study the effects of early initiation of alirocumab in addition to high intensity statin therapy in patients who have previously been treated with high intensity statins with poor response, who present with a type I (spontaneous) acute NSTEMI. Patients will be dosed with drug or placebo once during the first day of their hospital admission. Blood samples will be collected at baseline, 3 days and 14 days after randomization for biomarker testing. Particular attention will be paid to additional LDL lowering effects, as well as the effects on PCSK9 levels and inflammatory biomarkers. Safety and tolerability will be monitored with complete blood count + differential and complete metabolic panels at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Acute type I (spontaneous) NSTEMI defined as chest pain (or equivalent) with an onset of symptoms within 12 hours of presentation, a duration of >15 minutes, and elevated cardiac troponin I levels, with or without electrocardiographic changes [with the exclusion of ST elevation];
2. On medical therapy with high intensity statin prior to admission (either atorvastatin 40-80 mg or rosuvastatin 20-40 mg) as documented by hospital or pharmacy records and with known LDL cholesterol ≥70 mg/dL within the prior 12 months.

Exclusion Criteria:

1. Age <21 years of age
2. Inability to give informed consent
3. Previous, current or planned treatment with a PCSK9 inhibitor
4. Known history of loss of function of PCSK9 (genetic mutation or sequence variation)
5. Patient with homozygous familial hypercholesterolemia (clinically or by previous genotyping)
6. Recent (<14 days) or active use of immunosuppressive drugs (including but not limited to high-dose corticosteroids [>1mg/kg of prednisone equivalent], Tumor Necrosis Factor-α blockers, cyclosporine) not including non-steroidal antinflammatory drugs or corticosteroids used for IV dye allergy or corticosteroids used as replacement therapy for pituitary/adrenal disease with a stable regimen for at least 6 weeks prior to randomization (note: topical, intra-articular, nasal, inhaled, and ophthalmic steroid therapies are not considered "systemic" and are allowed);
7. Chronic auto-immune or auto-inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus);
8. History of cancer within the past 5 years, except for adequately treated basal cell skin cancer, squamous cell skin cancer, or in situ cervical cancer;
9. Known chronic hepatitis B or C infection (excluding patients with a positive antibody who were successfully treated or who have demonstrated no viral load);
10. Known human immunodeficiency virus infection.
11. Use of fibrates other than fenofibrate within 6 weeks of the screening visit.
12. Uncontrolled hypothyroidism. Note: patients on thyroid replacement therapy can be included if the dosage of thyroxin has been stable for at least 12 weeks prior to screening.
13. Known history of a hemorrhagic stroke.
14. Has been previously treated with at least 1 dose of alirocumab or any other anti-PCSK9 monoclonal antibody in other clinical studies.
15. Conditions/situations such as:

    1. Any clinically significant abnormality identified at the time of screening that in the judgment of the investigator or any sub-investigator would preclude safe completion of the study or constrain assessment of endpoints, such as major systemic diseases or patients with short life expectancy.
    2. Patients considered by the investigator or any sub-investigator to be inappropriate for this study for any reason:

    i. Those patients deemed unable to meet specific protocol requirements, such as scheduled visits.

    ii. Those patients the investigator deems unable to administer or tolerate long-term injections.

    c. Investigator or any sub-investigator, pharmacist, study coordinator, other study staff, or relative thereof directly involved in the conduct of the protocol.

    d. Presence of any other conditions (geographic or social), actual or anticipated, that the investigator feels would restrict or limit the patient's participation for the duration of the study.
16. Thyroid-stimulating hormone (TSH) < lower limit of normal (LLN) or > upper limit of normal (ULN); if TSH is abnormal due to controlled hypothyroidism (patient is on a stable dose of thyroid replacement therapy), the patient may be enrolled into the study;
17. Exclusion Criteria Related to the Active Comparator and/or Mandatory Background Therapies: All contraindications to the background therapies or warnings/precautions of use (when appropriate) as displayed in the respective national product labeling.
18. Exclusion Criteria Related to the Current Knowledge of Alirocumab

    1. Known hypersensitivity to monoclonal antibody therapeutics
    2. Pregnant or breastfeeding women
19. Women of childbearing potential who are not protected by highly effective method(s) of birth control throughout the entire duration of study treatment and for 10 weeks after the last dose of study drug and/or who are unwilling or unable to be tested for pregnancy.
20. Men capable of impregnating women who are not protected by highly effective method(s) of birth control and/or who are unwilling to use an effective contraceptive method throughout the entire duration of study treatment and for 10 weeks after the last dose of study drug.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to present the data promptly upon analysis as an abstract to a national meeting and/or a manuscript.

RESULTS

PARTICIPANT FLOW:
Groups:
- Alirocumab: Alirocumab (150 mg) will be administered by subcutaneous injection once, within the first day of the patient's diagnosis of NSTEMI. Patients will also receive an 80 mg dose of atorvastatin.
  alirocumab
- Placebo: Placebo (sterile saline) will be administered by subcutaneous injection once, within the first day of the patient's diagnosis of NSTEMI. Patients will also receive an 80 mg dose of atorvastatin.
  placebo
Period: Overall Study
Arm/Group | Alirocumab | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alirocumab | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [51 to 66] | 56 [48 to 65] | 59 [49 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 6 | 1 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
body mass index [Median (Inter-Quartile Range); unit: kilograms per meters squared] | 27.8 [24.2 to 36.8] | 31.9 [28.7 to 38.8] | 30.9 [25.5 to 37.4]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Low-density Lipoprotein (LDL) Cholesterol
Description: Placebo-corrected percentage change in calculated LDL cholesterol from baseline to day 14
Time Frame: baseline and 14 days
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Alirocumab | Placebo
Number analyzed (Participants) | 10 | 10
percent change | -73 [-83 to -56] | 2 [-12 to 11]
Statistical Analysis 1: Comparison: Alirocumab vs Placebo; Test type: Superiority; p < 0.01, ANOVA

2. Secondary Outcome: Change in Inflammatory Markers (hsCRP)
Description: Placebo-corrected percentage change in inflammatory markers (hsCRP) from baseline to 3 days
Time Frame: baseline to 3 days
Population: Research team was unable to collect samples from 2 Alirocumab participants.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Alirocumab | Placebo
Number analyzed (Participants) | 8 | 10
percent change | 58 [-27 to 82] | 55 [-25 to 161]
Statistical Analysis 1: Comparison: Alirocumab vs Placebo; Test type: Superiority; p > 0.20, ANOVA

3. Secondary Outcome: Change in Inflammatory Markers (hsCRP)
Description: Placebo-corrected Percentage Change in Inflammatory Markers (hsCRP) From Baseline to 14 Days
Time Frame: baseline to 14 days
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Alirocumab | Placebo
Number analyzed (Participants) | 10 | 10
percent change | -4 [-55 to 71] | -33 [-48 to 13]
Statistical Analysis 1: Comparison: Alirocumab vs Placebo; Test type: Superiority; p > 0.20, ANOVA

ADVERSE EVENTS:
Time Frame: From baseline to 14 days
Arm/Group | Alirocumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10 | 1/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alirocumab (N=10) | Placebo (N=10)
sepsis (Infections and infestations) | 0 (0) | 1 (1)
stroke (Nervous system disorders) | 1 (1) | 0 (0)
admission for heart failure (Cardiac disorders) | 2 (2) | 0 (0)
admission for unstable angina (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02938949/Prot_SAP_000.pdf